CLINICAL TRIAL: NCT02835261
Title: Impact of Sleep Restriction on Cardiometabolic Risk Factors in Pre vs Postmenopausal Women
Brief Title: Impact of Sleep Restriction in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Assistant Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AAAQ7638
Record Dates: First submitted 2016-06-21; First posted 2016-07-18 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Sleep; Cardiovascular Disease; Obesity
Keywords: Obesity; Metabolic Disorders
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Habitual Sleep (HS) (No Intervention): During the HS phase, participants will be asked to follow a fixed bedtime routine based on their screening sleep schedule.
- Sleep Restriction (SR) (Experimental): During the SR phase, participants will be asked to keep their habitual wake time constant but delay their bedtime to achieve a reduction of 1.5 h in total sleep time. A delay in bedtimes was chosen rather than advancing wakeup time because it most closely reflects differences in sleep timing behavior between short and normal sleepers.
  Interventions: Other: Sleep Restriction

INTERVENTIONS:
Other: Sleep Restriction — Mild sleep restriction (-1.5 h/night) over a period of 6 weeks
  Arms: Sleep Restriction (SR)

SUMMARY:
The overall goal of this project is to test the hypothesis that long-term, sustained sleep restriction (SR), in women, will lead to increased cardio-metabolic risk. This will be characterized by increases in visceral adiposity, unhealthy lifestyle behaviors (poor dietary quality and low physical activity) and cardio-metabolic risk factors (blood pressure, glucose intolerance) relative to habitual sleep (HS). The investigators expect these changes to be worse in pre- compared to post-menopausal women.

DETAILED DESCRIPTION:
This project is funded by the American Heart Association Go Red for Women Strategically Focused Research Network (SFRN). This SFRN includes two separate projects: Clinical Science Project (PI, St-Onge) and Basic Science Project (PI, Jelic). Women are enrolled in the Clinical Science project and given the option to enter the Basic Science project. Each project (clinical and basic) has its own separate primary and secondary outcomes. For the Clinical Science project, primary outcomes are glucose tolerance and ambulatory and office blood pressure; and secondary outcomes are body composition and circulating inflammatory markers. For the Basic Science project, the primary outcomes are flow mediated dilatation of the brachial artery (FMD) and secondary outcomes are endothelial cell oxidative stress and inflammation. The results of these two projects will be reported in separate and in combined publications.

This study will be a randomized, crossover, outpatient sleep restriction (SR) study with 2 phases of 6 weeks each, with a 6 week wash-out period between the phases. Sleep duration in each phase will be the participant's regular bed- and wake times during the habitual sleep (HS) phase and HS minus 1.5 hours in the SR phase. During the HS phase, participants will be asked to follow a fixed bedtime routine based on their screening sleep schedule. During the SR phase, participants will be asked to keep their habitual wake time constant but delay their bedtime to achieve a reduction of 1.5 hours in total sleep time.

On the first day of each study phase (baseline), participants will come to the research center in the morning after an overnight,12 hour fast. Participants will have anthropometric measurements taken and will then be taken to the department of Radiology to undergo magnetic resonance imaging (MRI) scanning to assess body composition. Flow-mediated dilatation will be performed in the Cardiovascular Ultrasound Laboratory followed by endothelial cell harvesting (Basic Science project). A sample of cells lining the blood vessel (forearm vein) will be taken to assess endothelial function. Women will undergo an oral glucose tolerance test (Clinical Science project). Blood samples will be taken for hormone measurements (insulin, cortisol). Participants will begin the fixed bedtime routine that night. These baseline measurements will be repeated at endpoint, 6 weeks later. Body weight and waist circumference will be measured weekly and fasting blood samples will be taken at weeks 3 and 4 during adherence check visits.

To verify that participants adhere to the sleep protocol, they will be asked to keep a sleep diary and wear an activity monitor 24 hours/day. Participants will wear an actigraph GT3X+ on their wrist, which will serve to track their sleep duration, sleep timing, and physical activity. Two weeks prior to randomization and during the washout period, participants will also wear the actigraph watch and keep a sleep diary to verify sleep duration and sleep-wake schedule. In addition to achieving an average sleep of 7-9 hours/night, by wrist actigraphy, participants will only be enrolled if they achieve 7 hours of sleep for at least 10 of the 14 nights of screening and have <4 nights with <6 hours of sleep. At the time of randomization, a urine pregnancy test and drug screen will be performed. Participants will be asked to abstain from caffeine and alcohol intake for 24 hours prior to the start. Between study phases, if participants have not returned to baseline sleep patterns within the 6 week washout period, an additional 2-4 week washout period will be provided. This washout length will ensure that women are in the same phase of their menstrual cycle at the start of each experimental phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years old
* All racial/ethnic groups
* Body mass index 18.5-34.9 kg/m2
* Sleep 7-9 h in bed/night with no daytime nap
* Normal scores on:

Pittsburgh Quality of Sleep Questionnaire Epworth Sleepiness Scale, Berlin Questionnaire, Sleep Disorders Inventory Questionnaire, Beck Depression Inventory, Composite Scale of Morningness/Eveningness, Three Factor Eating Questionnaire

Exclusion Criteria:

* Smokers (any cigarettes or ex-smoker <3 years)
* Neurological, medical or psychiatric disorder
* Diabetics
* Regular use of any medication or supplement
* Eating and/or sleep disorders
* Contraindications for MRI scanning
* Travel across time zones within 4 wk
* History of drug and alcohol abuse
* Shift worker (or rotating shift worker)
* Caffeine intake >300 mg/d
* Oral contraceptive use or hormone replacement therapy
* Heavy equipment operators
* Commercial long-distance drivers.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance | baseline to 6 weeks
  Oral glucose tolerance test
Change in blood pressure | baseline to 6 weeks
  24-hour ambulatory blood pressure; weekly office blood pressure
Flow-mediated dilatation | baseline to 6 weeks
  Endpoint FMD

SECONDARY OUTCOMES:
Change in Adiposity | baseline to 6 weeks
  Body composition measured by magnetic resonance imaging
Change in physical activity levels | baseline to 6 weeks
  Time in various behaviors: sedentary, light, moderate, moderate-to-vigorous physical activity
C-reactive protein | Weeks 0, 3, 4, and 6
  Inflammatory markers
Interleukin-6 | Weeks 0, 3, 4, and 6
  Inflammatory markers
Tumor necrosis factor | Weeks 0, 3, 4, and 6
  Inflammatory markers
T cell reactivity to viral loads | Weeks 0 and 6
  Immune markers
Cholesterol | Weeks 0 and 6
  Total, low-density, and high-density lipoprotein
Triglycerides | Weeks 0 and 6
  Lipidemia
Endothelial cell oxidative stress | Baseline to 6 weeks
  redox sensitive fluorogenic probe fluorescence intensity
Endothelial inflammation | baseline to 6 weeks
  NF-κB nuclear fluorescence area

OTHER OUTCOMES:
NIH Toolbox® for Assessment of Neurological and Behavioral Function (NIH Toolbox) | Weeks 0 and 6
  Neuro-behavioral assessments: cognition, motor, sensation raw scores

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University-New York Obesity Nutrition Research Center; Sanja Jelic, MD, Principal Investigator — Columbia University
Locations (1):
- New York Obesity Nutrition Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon study completion, after publication of main research aims.
Access Criteria: Contact PI directly

REFERENCES:
- [Background] Jackowska M, Steptoe A. Sleep and future cardiovascular risk: prospective analysis from the English Longitudinal Study of Ageing. Sleep Med. 2015 Jun;16(6):768-74. doi: 10.1016/j.sleep.2015.02.530. Epub 2015 Mar 9. PMID 25934538
- [Background] Wu MC, Yang YC, Wu JS, Wang RH, Lu FH, Chang CJ. Short sleep duration associated with a higher prevalence of metabolic syndrome in an apparently healthy population. Prev Med. 2012 Oct;55(4):305-309. doi: 10.1016/j.ypmed.2012.07.013. Epub 2012 Jul 27. PMID 22846501
- [Background] Ohkuma T, Fujii H, Iwase M, Ogata-Kaizu S, Ide H, Kikuchi Y, Idewaki Y, Jodai T, Hirakawa Y, Nakamura U, Kitazono T. U-shaped association of sleep duration with metabolic syndrome and insulin resistance in patients with type 2 diabetes: the Fukuoka Diabetes Registry. Metabolism. 2014 Apr;63(4):484-91. doi: 10.1016/j.metabol.2013.12.001. Epub 2013 Dec 7. PMID 24411997
- [Background] Chaput JP, McNeil J, Despres JP, Bouchard C, Tremblay A. Seven to eight hours of sleep a night is associated with a lower prevalence of the metabolic syndrome and reduced overall cardiometabolic risk in adults. PLoS One. 2013 Sep 5;8(9):e72832. doi: 10.1371/journal.pone.0072832. eCollection 2013. PMID 24039808
- [Background] Hall MH, Muldoon MF, Jennings JR, Buysse DJ, Flory JD, Manuck SB. Self-reported sleep duration is associated with the metabolic syndrome in midlife adults. Sleep. 2008 May;31(5):635-43. doi: 10.1093/sleep/31.5.635. PMID 18517034
- [Background] Chaput JP, McNeil J, Despres JP, Bouchard C, Tremblay A. Short sleep duration as a risk factor for the development of the metabolic syndrome in adults. Prev Med. 2013 Dec;57(6):872-7. doi: 10.1016/j.ypmed.2013.09.022. Epub 2013 Oct 5. PMID 24099879
- [Background] Cappuccio FP, Taggart FM, Kandala NB, Currie A, Peile E, Stranges S, Miller MA. Meta-analysis of short sleep duration and obesity in children and adults. Sleep. 2008 May;31(5):619-26. doi: 10.1093/sleep/31.5.619. PMID 18517032
- [Background] Redline S, Foody J. Sleep disturbances: time to join the top 10 potentially modifiable cardiovascular risk factors? Circulation. 2011 Nov 8;124(19):2049-51. doi: 10.1161/CIRCULATIONAHA.111.062190. No abstract available. PMID 22064955
- [Background] Robertson MD, Russell-Jones D, Umpleby AM, Dijk DJ. Effects of three weeks of mild sleep restriction implemented in the home environment on multiple metabolic and endocrine markers in healthy young men. Metabolism. 2013 Feb;62(2):204-11. doi: 10.1016/j.metabol.2012.07.016. Epub 2012 Sep 15. PMID 22985906
- [Background] Hoevenaar-Blom MP, Spijkerman AM, Kromhout D, Verschuren WM. Sufficient sleep duration contributes to lower cardiovascular disease risk in addition to four traditional lifestyle factors: the MORGEN study. Eur J Prev Cardiol. 2014 Nov;21(11):1367-75. doi: 10.1177/2047487313493057. Epub 2013 Jul 3. PMID 23823570
- [Background] Ford ES. Habitual sleep duration and predicted 10-year cardiovascular risk using the pooled cohort risk equations among US adults. J Am Heart Assoc. 2014 Dec 2;3(6):e001454. doi: 10.1161/JAHA.114.001454. PMID 25468656
- [Background] Canivet C, Nilsson PM, Lindeberg SI, Karasek R, Ostergren PO. Insomnia increases risk for cardiovascular events in women and in men with low socioeconomic status: a longitudinal, register-based study. J Psychosom Res. 2014 Apr;76(4):292-9. doi: 10.1016/j.jpsychores.2014.02.001. Epub 2014 Feb 11. PMID 24630179
- [Background] Sands-Lincoln M, Loucks EB, Lu B, Carskadon MA, Sharkey K, Stefanick ML, Ockene J, Shah N, Hairston KG, Robinson JG, Limacher M, Hale L, Eaton CB. Sleep duration, insomnia, and coronary heart disease among postmenopausal women in the Women's Health Initiative. J Womens Health (Larchmt). 2013 Jun;22(6):477-86. doi: 10.1089/jwh.2012.3918. Epub 2013 May 7. PMID 23651054
- [Background] Cappuccio FP, Cooper D, D'Elia L, Strazzullo P, Miller MA. Sleep duration predicts cardiovascular outcomes: a systematic review and meta-analysis of prospective studies. Eur Heart J. 2011 Jun;32(12):1484-92. doi: 10.1093/eurheartj/ehr007. Epub 2011 Feb 7. PMID 21300732
- [Background] Cappuccio FP, Stranges S, Kandala NB, Miller MA, Taggart FM, Kumari M, Ferrie JE, Shipley MJ, Brunner EJ, Marmot MG. Gender-specific associations of short sleep duration with prevalent and incident hypertension: the Whitehall II Study. Hypertension. 2007 Oct;50(4):693-700. doi: 10.1161/HYPERTENSIONAHA.107.095471. Epub 2007 Sep 4. PMID 17785629
- [Background] Stranges S, Dorn JM, Cappuccio FP, Donahue RP, Rafalson LB, Hovey KM, Freudenheim JL, Kandala NB, Miller MA, Trevisan M. A population-based study of reduced sleep duration and hypertension: the strongest association may be in premenopausal women. J Hypertens. 2010 May;28(5):896-902. doi: 10.1097/HJH.0b013e328335d076. PMID 20040890
- [Background] Gangwisch JE, Feskanich D, Malaspina D, Shen S, Forman JP. Sleep duration and risk for hypertension in women: results from the nurses' health study. Am J Hypertens. 2013 Jul;26(7):903-11. doi: 10.1093/ajh/hpt044. Epub 2013 Apr 4. PMID 23564028
- [Background] Choi JK, Kim MY, Kim JK, Park JK, Oh SS, Koh SB, Eom A. Association between short sleep duration and high incidence of metabolic syndrome in midlife women. Tohoku J Exp Med. 2011 Nov;225(3):187-93. doi: 10.1620/tjem.225.187. PMID 22001675
- [Background] Miller MA, Kandala NB, Kivimaki M, Kumari M, Brunner EJ, Lowe GD, Marmot MG, Cappuccio FP. Gender differences in the cross-sectional relationships between sleep duration and markers of inflammation: Whitehall II study. Sleep. 2009 Jul;32(7):857-64. PMID 19639748
- [Background] Matthews KA, Zheng H, Kravitz HM, Sowers M, Bromberger JT, Buysse DJ, Owens JF, Sanders M, Hall M. Are inflammatory and coagulation biomarkers related to sleep characteristics in mid-life women?: Study of Women's Health across the Nation sleep study. Sleep. 2010 Dec;33(12):1649-55. doi: 10.1093/sleep/33.12.1649. PMID 21120127
- [Background] St-Onge MP, Perumean-Chaney S, Desmond R, Lewis CE, Yan LL, Person SD, Allison DB. Gender Differences in the Association between Sleep Duration and Body Composition: The Cardia Study. Int J Endocrinol. 2010;2010:726071. doi: 10.1155/2010/726071. Epub 2009 Nov 12. PMID 20049158
- [Background] Mezick EJ, Wing RR, McCaffery JM. Associations of self-reported and actigraphy-assessed sleep characteristics with body mass index and waist circumference in adults: moderation by gender. Sleep Med. 2014 Jan;15(1):64-70. doi: 10.1016/j.sleep.2013.08.784. Epub 2013 Oct 14. PMID 24239499
- [Background] Bosy-Westphal A, Hinrichs S, Jauch-Chara K, Hitze B, Later W, Wilms B, Settler U, Peters A, Kiosz D, Muller MJ. Influence of partial sleep deprivation on energy balance and insulin sensitivity in healthy women. Obes Facts. 2008;1(5):266-73. doi: 10.1159/000158874. Epub 2008 Oct 23. PMID 20054188
- [Background] Markwald RR, Melanson EL, Smith MR, Higgins J, Perreault L, Eckel RH, Wright KP Jr. Impact of insufficient sleep on total daily energy expenditure, food intake, and weight gain. Proc Natl Acad Sci U S A. 2013 Apr 2;110(14):5695-700. doi: 10.1073/pnas.1216951110. Epub 2013 Mar 11. PMID 23479616
- [Background] Spaeth AM, Dinges DF, Goel N. Effects of Experimental Sleep Restriction on Weight Gain, Caloric Intake, and Meal Timing in Healthy Adults. Sleep. 2013 Jul 1;36(7):981-990. doi: 10.5665/sleep.2792. PMID 23814334
- [Background] Nedeltcheva AV, Kilkus JM, Imperial J, Kasza K, Schoeller DA, Penev PD. Sleep curtailment is accompanied by increased intake of calories from snacks. Am J Clin Nutr. 2009 Jan;89(1):126-33. doi: 10.3945/ajcn.2008.26574. Epub 2008 Dec 3. PMID 19056602
- [Background] St-Onge MP, Roberts AL, Chen J, Kelleman M, O'Keeffe M, RoyChoudhury A, Jones PJ. Short sleep duration increases energy intakes but does not change energy expenditure in normal-weight individuals. Am J Clin Nutr. 2011 Aug;94(2):410-6. doi: 10.3945/ajcn.111.013904. Epub 2011 Jun 29. PMID 21715510
- [Background] Shechter A, Rising R, Albu JB, St-Onge MP. Experimental sleep curtailment causes wake-dependent increases in 24-h energy expenditure as measured by whole-room indirect calorimetry. Am J Clin Nutr. 2013 Dec;98(6):1433-9. doi: 10.3945/ajcn.113.069427. Epub 2013 Oct 2. PMID 24088722
- [Background] Haack M, Sanchez E, Mullington JM. Elevated inflammatory markers in response to prolonged sleep restriction are associated with increased pain experience in healthy volunteers. Sleep. 2007 Sep;30(9):1145-52. doi: 10.1093/sleep/30.9.1145. PMID 17910386
- [Background] van Leeuwen WM, Lehto M, Karisola P, Lindholm H, Luukkonen R, Sallinen M, Harma M, Porkka-Heiskanen T, Alenius H. Sleep restriction increases the risk of developing cardiovascular diseases by augmenting proinflammatory responses through IL-17 and CRP. PLoS One. 2009;4(2):e4589. doi: 10.1371/journal.pone.0004589. Epub 2009 Feb 25. PMID 19240794
- [Background] Meier-Ewert HK, Ridker PM, Rifai N, Regan MM, Price NJ, Dinges DF, Mullington JM. Effect of sleep loss on C-reactive protein, an inflammatory marker of cardiovascular risk. J Am Coll Cardiol. 2004 Feb 18;43(4):678-83. doi: 10.1016/j.jacc.2003.07.050. PMID 14975482
- [Background] Frey DJ, Fleshner M, Wright KP Jr. The effects of 40 hours of total sleep deprivation on inflammatory markers in healthy young adults. Brain Behav Immun. 2007 Nov;21(8):1050-7. doi: 10.1016/j.bbi.2007.04.003. Epub 2007 May 23. PMID 17524614
- [Background] Kerkhofs M, Boudjeltia KZ, Stenuit P, Brohee D, Cauchie P, Vanhaeverbeek M. Sleep restriction increases blood neutrophils, total cholesterol and low density lipoprotein cholesterol in postmenopausal women: A preliminary study. Maturitas. 2007 Feb 20;56(2):212-5. doi: 10.1016/j.maturitas.2006.07.007. Epub 2006 Sep 1. PMID 16950577
- [Background] O'Keeffe M, Roberts AL, Kelleman M, Roychoudhury A, St-Onge MP. No effects of short-term sleep restriction, in a controlled feeding setting, on lipid profiles in normal-weight adults. J Sleep Res. 2013 Dec;22(6):717-20. doi: 10.1111/jsr.12060. Epub 2013 May 20. PMID 23682639
- [Background] Spiegel K, Leproult R, Van Cauter E. Impact of sleep debt on metabolic and endocrine function. Lancet. 1999 Oct 23;354(9188):1435-9. doi: 10.1016/S0140-6736(99)01376-8. PMID 10543671
- [Background] Spiegel K, Knutson K, Leproult R, Tasali E, Van Cauter E. Sleep loss: a novel risk factor for insulin resistance and Type 2 diabetes. J Appl Physiol (1985). 2005 Nov;99(5):2008-19. doi: 10.1152/japplphysiol.00660.2005. PMID 16227462
- [Background] Van Cauter E, Spiegel K, Tasali E, Leproult R. Metabolic consequences of sleep and sleep loss. Sleep Med. 2008 Sep;9 Suppl 1(0 1):S23-8. doi: 10.1016/S1389-9457(08)70013-3. PMID 18929315
- [Background] Donga E, van Dijk M, van Dijk JG, Biermasz NR, Lammers GJ, van Kralingen KW, Corssmit EP, Romijn JA. A single night of partial sleep deprivation induces insulin resistance in multiple metabolic pathways in healthy subjects. J Clin Endocrinol Metab. 2010 Jun;95(6):2963-8. doi: 10.1210/jc.2009-2430. Epub 2010 Apr 6. PMID 20371664
- [Background] Schmid SM, Hallschmid M, Jauch-Chara K, Wilms B, Lehnert H, Born J, Schultes B. Disturbed glucoregulatory response to food intake after moderate sleep restriction. Sleep. 2011 Mar 1;34(3):371-7. doi: 10.1093/sleep/34.3.371. PMID 21358855
- [Background] Buxton OM, Pavlova M, Reid EW, Wang W, Simonson DC, Adler GK. Sleep restriction for 1 week reduces insulin sensitivity in healthy men. Diabetes. 2010 Sep;59(9):2126-33. doi: 10.2337/db09-0699. Epub 2010 Jun 28. PMID 20585000
- [Background] Nedeltcheva AV, Kessler L, Imperial J, Penev PD. Exposure to recurrent sleep restriction in the setting of high caloric intake and physical inactivity results in increased insulin resistance and reduced glucose tolerance. J Clin Endocrinol Metab. 2009 Sep;94(9):3242-50. doi: 10.1210/jc.2009-0483. Epub 2009 Jun 30. PMID 19567526
- [Background] Mosca M, Aggarwal B. Sleep duration, snoring habits, and cardiovascular disease risk factors in an ethnically diverse population. J Cardiovasc Nurs. 2012 May-Jun;27(3):263-9. doi: 10.1097/JCN.0b013e31821e7ad1. PMID 21743341
- [Background] Prather AA, Epel ES, Cohen BE, Neylan TC, Whooley MA. Gender differences in the prospective associations of self-reported sleep quality with biomarkers of systemic inflammation and coagulation: findings from the Heart and Soul Study. J Psychiatr Res. 2013 Sep;47(9):1228-35. doi: 10.1016/j.jpsychires.2013.05.004. Epub 2013 Jun 5. PMID 23746737
- [Background] St-Onge MP, O'Keeffe M, Roberts AL, RoyChoudhury A, Laferrere B. Short sleep duration, glucose dysregulation and hormonal regulation of appetite in men and women. Sleep. 2012 Nov 1;35(11):1503-10. doi: 10.5665/sleep.2198. PMID 23115399
- [Background] Shechter A, Rising R, Wolfe S, Albu JB, St-Onge MP. Postprandial thermogenesis and substrate oxidation are unaffected by sleep restriction. Int J Obes (Lond). 2014 Sep;38(9):1153-8. doi: 10.1038/ijo.2013.239. Epub 2013 Dec 19. PMID 24352294
- [Background] St-Onge MP, Shechter A, Shlisky J, Tam CS, Gao S, Ravussin E, Butler AA. Fasting plasma adropin concentrations correlate with fat consumption in human females. Obesity (Silver Spring). 2014 Apr;22(4):1056-63. doi: 10.1002/oby.20631. Epub 2013 Oct 17. PMID 24115373
- [Background] St-Onge MP, Wolfe S, Sy M, Shechter A, Hirsch J. Sleep restriction increases the neuronal response to unhealthy food in normal-weight individuals. Int J Obes (Lond). 2014 Mar;38(3):411-6. doi: 10.1038/ijo.2013.114. Epub 2013 Jun 19. PMID 23779051
- [Background] Shechter A, O'Keeffe M, Roberts AL, Zammit GK, RoyChoudhury A, St-Onge MP. Alterations in sleep architecture in response to experimental sleep curtailment are associated with signs of positive energy balance. Am J Physiol Regul Integr Comp Physiol. 2012 Nov 1;303(9):R883-9. doi: 10.1152/ajpregu.00222.2012. Epub 2012 Sep 12. PMID 22972835
- [Background] St-Onge MP, McReynolds A, Trivedi ZB, Roberts AL, Sy M, Hirsch J. Sleep restriction leads to increased activation of brain regions sensitive to food stimuli. Am J Clin Nutr. 2012 Apr;95(4):818-24. doi: 10.3945/ajcn.111.027383. Epub 2012 Feb 22. PMID 22357722
- [Background] St-Onge MP, Roberts A, Shechter A, Choudhury AR. Fiber and Saturated Fat Are Associated with Sleep Arousals and Slow Wave Sleep. J Clin Sleep Med. 2016 Jan;12(1):19-24. doi: 10.5664/jcsm.5384. PMID 26156950
- [Background] St-Onge MP. The role of sleep duration in the regulation of energy balance: effects on energy intakes and expenditure. J Clin Sleep Med. 2013 Jan 15;9(1):73-80. doi: 10.5664/jcsm.2348. PMID 23319909
- [Background] Shechter A, Grandner MA, St-Onge MP. The Role of Sleep in the Control of Food Intake. Am J Lifestyle Med. 2014 Nov 1;8(6):371-374. doi: 10.1177/1559827614545315. Epub 2014 Aug 6. PMID 27065757
- [Background] St-Onge MP, Shechter A. Sleep disturbances, body fat distribution, food intake and/or energy expenditure: pathophysiological aspects. Horm Mol Biol Clin Investig. 2014 Jan;17(1):29-37. doi: 10.1515/hmbci-2013-0066. PMID 25372728
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Douglass AB, Bornstein R, Nino-Murcia G, Keenan S, Miles L, Zarcone VP Jr, Guilleminault C, Dement WC. The Sleep Disorders Questionnaire. I: Creation and multivariate structure of SDQ. Sleep. 1994 Mar;17(2):160-7. doi: 10.1093/sleep/17.2.160. PMID 8036370
- [Background] Arnau RC, Meagher MW, Norris MP, Bramson R. Psychometric evaluation of the Beck Depression Inventory-II with primary care medical patients. Health Psychol. 2001 Mar;20(2):112-9. doi: 10.1037//0278-6133.20.2.112. PMID 11315728
- [Background] Smith CS, Reilly C, Midkiff K. Evaluation of three circadian rhythm questionnaires with suggestions for an improved measure of morningness. J Appl Psychol. 1989 Oct;74(5):728-38. doi: 10.1037/0021-9010.74.5.728. PMID 2793773
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Silva GE, Goodwin JL, Sherrill DL, Arnold JL, Bootzin RR, Smith T, Walsleben JA, Baldwin CM, Quan SF. Relationship between reported and measured sleep times: the sleep heart health study (SHHS). J Clin Sleep Med. 2007 Oct 15;3(6):622-30. PMID 17993045
- [Background] Basner M, Dinges DF. Dubious bargain: trading sleep for Leno and Letterman. Sleep. 2009 Jun;32(6):747-52. doi: 10.1093/sleep/32.6.747. PMID 19544750
- [Background] Asarnow LD, McGlinchey E, Harvey AG. The effects of bedtime and sleep duration on academic and emotional outcomes in a nationally representative sample of adolescents. J Adolesc Health. 2014 Mar;54(3):350-6. doi: 10.1016/j.jadohealth.2013.09.004. Epub 2013 Nov 10. PMID 24225447
- [Background] Reid KJ, Santostasi G, Baron KG, Wilson J, Kang J, Zee PC. Timing and intensity of light correlate with body weight in adults. PLoS One. 2014 Apr 2;9(4):e92251. doi: 10.1371/journal.pone.0092251. eCollection 2014. PMID 24694994
- [Background] Spaeth AM, Dinges DF, Goel N. Sex and race differences in caloric intake during sleep restriction in healthy adults. Am J Clin Nutr. 2014 Aug;100(2):559-66. doi: 10.3945/ajcn.114.086579. Epub 2014 Jun 25. PMID 24965304
- [Background] Shen W, Chen J, Kwak S, Punyanitya M, Heymsfield SB. Between-slice intervals in quantification of adipose tissue and muscle in children. Int J Pediatr Obes. 2011 Apr;6(2):149-56. doi: 10.3109/17477166.2010.486833. Epub 2010 Jun 7. PMID 20528126
- [Background] Gallagher D, Kuznia P, Heshka S, Albu J, Heymsfield SB, Goodpaster B, Visser M, Harris TB. Adipose tissue in muscle: a novel depot similar in size to visceral adipose tissue. Am J Clin Nutr. 2005 Apr;81(4):903-10. doi: 10.1093/ajcn/81.4.903. PMID 15817870
- [Background] St-Onge MP, Bourque C, Jones PJ, Ross R, Parsons WE. Medium- versus long-chain triglycerides for 27 days increases fat oxidation and energy expenditure without resulting in changes in body composition in overweight women. Int J Obes Relat Metab Disord. 2003 Jan;27(1):95-102. doi: 10.1038/sj.ijo.0802169. PMID 12532160
- [Background] St-Onge MP, Ross R, Parsons WD, Jones PJ. Medium-chain triglycerides increase energy expenditure and decrease adiposity in overweight men. Obes Res. 2003 Mar;11(3):395-402. doi: 10.1038/oby.2003.53. PMID 12634436
- [Background] Shen W, Chen J, Gantz M, Velasquez G, Punyanitya M, Heymsfield SB. A single MRI slice does not accurately predict visceral and subcutaneous adipose tissue changes during weight loss. Obesity (Silver Spring). 2012 Dec;20(12):2458-63. doi: 10.1038/oby.2012.168. Epub 2012 Jun 25. PMID 22728693
- [Background] Dhurandhar NV, Schoeller D, Brown AW, Heymsfield SB, Thomas D, Sorensen TI, Speakman JR, Jeansonne M, Allison DB; Energy Balance Measurement Working Group. Energy balance measurement: when something is not better than nothing. Int J Obes (Lond). 2015 Jul;39(7):1109-13. doi: 10.1038/ijo.2014.199. Epub 2014 Nov 13. PMID 25394308
- [Background] Berk ES, Kovera AJ, Boozer CN, Pi-Sunyer FX, Albu JB. Metabolic inflexibility in substrate use is present in African-American but not Caucasian healthy, premenopausal, nondiabetic women. J Clin Endocrinol Metab. 2006 Oct;91(10):4099-106. doi: 10.1210/jc.2005-2411. Epub 2006 Jul 25. PMID 16868062
- [Result] St-Onge MP, Campbell A, Aggarwal B, Taylor JL, Spruill TM, RoyChoudhury A. Mild sleep restriction increases 24-hour ambulatory blood pressure in premenopausal women with no indication of mediation by psychological effects. Am Heart J. 2020 May;223:12-22. doi: 10.1016/j.ahj.2020.02.006. Epub 2020 Feb 8. PMID 32135337
- [Result] St-Onge MP, Campbell A, Salazar I, Pizinger T, Liao M, Aggarwal B. Information on Bedtimes and Wake Times Improves the Relation Between Self-Reported and Objective Assessments of Sleep in Adults. J Clin Sleep Med. 2019 Jul 15;15(7):1031-1036. doi: 10.5664/jcsm.7888. PMID 31383241
- [Result] St-Onge MP, Campbell A, Zuraikat F, Cheng B, Shah R, Berger JS, Sampogna RV, Jelic S. Impact of change in bedtime variability on body composition and inflammation: secondary findings from the Go Red for Women Strategically Focused Research Network. Int J Obes (Lond). 2020 Aug;44(8):1803-1806. doi: 10.1038/s41366-020-0555-1. Epub 2020 Mar 5. PMID 32132641
- [Result] Aggarwal B, Makarem N, Shah R, Emin M, Wei Y, St-Onge MP, Jelic S. Effects of Inadequate Sleep on Blood Pressure and Endothelial Inflammation in Women: Findings From the American Heart Association Go Red for Women Strategically Focused Research Network. J Am Heart Assoc. 2018 Jun 9;7(12):e008590. doi: 10.1161/JAHA.118.008590. PMID 29886425
- [Result] Makarem N, Zuraikat FM, Scaccia SE, RoyChoudhury A, St-Onge MP. Sustained Mild Sleep Restriction Increases Blood Pressure in Women: An Update From the American Heart Association Go Red for Women Strategically Focused Research Network. Hypertension. 2021 May 5;77(5):e50-e52. doi: 10.1161/HYPERTENSIONAHA.120.16370. Epub 2021 Mar 29. No abstract available. PMID 33775114
- [Result] Barragan R, Zuraikat FM, Tam V, Scaccia S, Cochran J, Li S, Cheng B, St-Onge MP. Actigraphy-Derived Sleep Is Associated with Eating Behavior Characteristics. Nutrients. 2021 Mar 5;13(3):852. doi: 10.3390/nu13030852. PMID 33807690
- [Result] St-Onge MP, Aggarwal B, Allison MA, Berger JS, Castaneda SF, Catov J, Hochman JS, Hubel CA, Jelic S, Kass DA, Makarem N, Michos ED, Mosca L, Ouyang P, Park C, Post WS, Powers RW, Reynolds HR, Sears DD, Shah SJ, Sharma K, Spruill T, Talavera GA, Vaidya D. Go Red for Women Strategically Focused Research Network: Summary of Findings and Network Outcomes. J Am Heart Assoc. 2021 Feb;10(5):e019519. doi: 10.1161/JAHA.120.019519. Epub 2021 Feb 23. PMID 33619972
- [Derived] Petrov ME, Zuraikat FM, Cheng B, Aggarwal B, Jelic S, Laferrere B, St-Onge MP. Impact of sleep restriction on biomarkers of thyroid function: Two pooled randomized trials. Sleep Med. 2024 Dec;124:606-612. doi: 10.1016/j.sleep.2024.10.035. Epub 2024 Oct 30. PMID 39488926
- [Derived] Zimmerman ME, Benasi G, Hale C, Yeung LK, Cochran J, Brickman AM, St-Onge MP. The effects of insufficient sleep and adequate sleep on cognitive function in healthy adults. Sleep Health. 2024 Apr;10(2):229-236. doi: 10.1016/j.sleh.2023.11.011. Epub 2024 Jan 16. PMID 38233280
- [Derived] Barragan R, Zuraikat FM, Cheng B, Scaccia SE, Cochran J, Aggarwal B, Jelic S, St-Onge MP. Paradoxical Effects of Prolonged Insufficient Sleep on Lipid Profile: A Pooled Analysis of 2 Randomized Trials. J Am Heart Assoc. 2023 Oct 17;12(20):e032078. doi: 10.1161/JAHA.123.032078. Epub 2023 Oct 10. PMID 37815115
- [Derived] Shah R, Shah VK, Emin M, Gao S, Sampogna RV, Aggarwal B, Chang A, St-Onge MP, Malik V, Wang J, Wei Y, Jelic S. Mild sleep restriction increases endothelial oxidative stress in female persons. Sci Rep. 2023 Sep 16;13(1):15360. doi: 10.1038/s41598-023-42758-y. PMID 37717072
- [Derived] Barragan R, Zuraikat FM, Tam V, RoyChoudhury A, St-Onge MP. Changes in eating patterns in response to chronic insufficient sleep and their associations with diet quality: a randomized trial. J Clin Sleep Med. 2023 Nov 1;19(11):1867-1875. doi: 10.5664/jcsm.10696. PMID 37409467

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02835261/Prot_SAP_000.pdf